CLINICAL TRIAL: NCT06034951
Title: Acceptability (including Gastrointestinal Tolerance and Compliance) of a High Energy, Adult Enteral Formula with Food-derived Ingredients.
Brief Title: Acceptability and Tolerance Study of a High Energy Tube Feed with Food Derived Ingredients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Compleat002
Record Dates: First submitted 2023-08-22; First posted 2023-09-13 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-04

CONDITIONS: Tolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients well established on tube feeds will act as their own control (Other): These patients will switch from current to new tube feed to assess acceptability and tolerance
  Interventions: Dietary Supplement: Compleat 1.5 HP

INTERVENTIONS:
Dietary Supplement: Compleat 1.5 HP — Patients well established and stable on an enteral tube feed. This group will act as their own controls and switched to the new tube feed.

SUMMARY:
Enterally fed adults and children who are assessed by the dietitian as requiring an adult high-energy, fibre-containing enteral formula will be recruited. Data from 15 participants are required in order to submit an application to the Advisory Committee on Borderline Substances (ACBS) for product registration.

DETAILED DESCRIPTION:
To evaluate the acceptability (including gastrointestinal tolerance and compliance) of a high energy, adult enteral formula with food-derived ingredients.This is a single arm, prospective, multi-centre study to evaluate the gastrointestinal tolerance and compliance over a 14-day period with the new tube feed.

Participants or their caregivers will be provided with 14-day supply of the new tube feed and will be asked to complete a daily diary and short questionnaire to record information allowing assessment of the following:

* Gastrointestinal tolerance
* Compliance with prescribed feed volume

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring an enteral tube feed (taking > 60% of energy needs from their feeding tube) as part of their dietary management for disease related malnutrition

  * Children 15 years and over
  * Adults and children requiring an adult high-energy and fibre-containing formula, as assessed by the dietitian.
  * Patients well-established and stable on enteral feeding.
  * Willingly given, written, informed consent from patient or consultee
  * Willingly given, written assent (if appropriate).

Exclusion Criteria:

* Inability to comply with the study protocol, in the opinion of the investigator

  * Children under 15 years of age
  * Patients receiving mechanical ventilation, sedation or inotropic support
  * Patients on total parenteral nutrition
  * Known food allergies to any ingredients (see ingredients list) or galactosaemia
  * Patients with significant renal or hepatic impairment
  * Patients with planned changes to medication or treatments during the study period which may alter gastrointestinal function (e.g. chemotherapy). Changes in medications or nutritional products during the study intervention must be documented.
  * Participation in another interventional study within 2 weeks of this study.
  * Patients with a clinical indication for a low fibre or fibre free diet as advised by the healthcare team.
  * Patients with known or suspected ileus or mechanical bowel obstruction

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-05-24 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Daily patient diaries | 14 days
  Daily monitor of gastrointestinal tolerance using questionnaire on increase, decrease or no change
Daily formula intake | 14 days
  mL per day

CONTACTS AND LOCATIONS:
Overall Officials: Martha Van Der Linde, Principal Investigator — Community Paediatric Dietitian Worcestershire North Nutrition and Dietetic Hastings Way, Worcester. UK; Amy Carter, Principal Investigator — The Walton Centre NHS Foundation Trust, Liverpool UK; Sam Ogundere, Principal Investigator — Lewisham and Greenwich NHS Trust London UK; Adrian Gilson, Principal Investigator — Newham General Hospital London UK
Locations (1):
- Martha Van Der Linde, Worcester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
will upload the data as it becomes available